CLINICAL TRIAL: NCT00275405
Title: Effect of Garlic Oil Macerate on Inflammatory Mediators in Healthy Normal Weight and Obese Subjects.
Brief Title: Effect of Garlic on Inflammatory Mediators
Status: Suspended | Phase: Phase 4 | Type: Interventional
Why Stopped: Results inconclusive
Sponsor: Albany Medical College (Other)
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: Ajoene
Record Dates: First submitted 2006-01-10; First posted 2006-01-12 (Estimated); Last update posted 2007-03-20 (Estimated); Status verified 2007-03

CONDITIONS: Healthy
Keywords: Effects of Garlic

INTERVENTIONS:
Drug: Garlic Oil Macerate

SUMMARY:
This research will investigate the effect of garlic oil extract when added to daily diet on inflammatory mediators and blood clotting activation.

DETAILED DESCRIPTION:
To investigate the pharmacokinetics of one of the garlic oil macerate, Ajoene, the anti-inflammatory effect of garlic oil macerate on the pro-inflammatory transcription factor NF-kB, it's activating proteins, including IkB, IkB Kinases a and B (IKKa and IKKB) and the pro-inflammatory NF-kB-regulated proteins, c-reactive protein (CRP), tumor necrosis factor-alpha (TNF-a), soluble intercellular adhesion molecule-1 (sICAM-1), soluble vascular cell adhesion molecule-1 (sVCAM-1), matrix metalloproteinase-9 (MMP-9), plasminogen activated protein-1 (PAI-1)and the effect of garlic oil macerate intake on platelet activation in normal subjects.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Normal subjects with BMI <25, obese subjects with BMI >30
* Subjects who have consented to adhere to the diet, regular weekly visits, and blood draws.

Exclusion Criteria:

* Subjects on any antioxidant medication.
* Patient on non-steroidal anti-inflammatory drug.
* On any agent with antioxidant properties.
* History of drug or alcohol abuse.
* Any life threatening disease.
* On any agent with significant antioxidant properties.
* Taking garlic extracts in the diet regularly.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34
Dates: Start 2006-04; Study Completion 2007-03 (Estimated)

PRIMARY OUTCOMES:
1. To examine the pharmacokinetics of the garlic oil macerate.

SECONDARY OUTCOMES:
2. To examine the effect of garlic oil macerate on inflammatory mechanisms at the cellular and molecular level.

CONTACTS AND LOCATIONS:
Overall Officials: Howard S Smith, MD, Principal Investigator — Albany Medical College; Shaker A Mousa, PhD, Principal Investigator — Albany College of Pharmacy; Ahmad Aljada, PhD, Principal Investigator — Albany College of Pharmacy
Locations (1):
- Albany Medical Center, Albany, New York, United States